CLINICAL TRIAL: NCT02227498
Title: Argus II Retinal Prosthesis System Dry AMD Feasibility Study Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Sight Medical Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-04-01
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Effect of Argus II on Functional Vision (Experimental): All subjects enrolled in the study will be implanted with the Argus II Retinal Prosthesis. To evaluate safety and effectiveness of Argus II on visual function.
  Interventions: Device: Effect of Argus II on Functional Vision

INTERVENTIONS:
Device: Effect of Argus II on Functional Vision — To evaluate the safety and effectiveness of the Argus II Retinal Prosthesis in subjects with AMD.

SUMMARY:
The purpose of this study is to test the Argus II Retinal Prosthesis System in patients with severe age-related macular degeneration (AMD). The Argus II System has already been studied in completely blind patients with retinitis pigmentosa (RP). In RP patients, some cells of the retina are irrevocably damaged and the Argus II System has been found to restore some basic visual function. On these grounds, the device has received authorization for use on the European market (the CE certification) in 2011.

DETAILED DESCRIPTION:
In this study, 5 subjects with severe dry AMD who are legally blind will be implanted with the Argus II System. The study will evaluate the safety of the device and surgery, as well as functioning of the system and the extent of any restored vision. Each subject will be followed for 3 years, with their eye health and visual function tested at multiple time points.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must consent to participate in the study;
2. Subject must be between 25 and 85 years of age;
3. Subject must be diagnosed with dry AMD (i.e., evidence of drusen and hyperplasia of the RPE in the eye with geographic atrophy secondary to dry AMD);
4. Severely sight impaired and meets the following additional criteria:

   1. Visual acuity of logMAR 1.0 (6/60) or worse in both eyes as measured by ETDRS;
   2. Hand motion or worse central vision in the eye to be implanted, as measured with a pinhole occluder;
   3. Geographic atrophy (confirmed by Fundus Autofluorescence) and central scotoma (confirmed by microperimetry) in the central 20° or more;
5. Subject must be pseudophakic with an IOL successfully implanted in the study eye at least 2 weeks before baseline testing, or aphakic with a clear capsule. If applicable, posterior laser capsulotomy may be performed 2 weeks before baseline testing is performed;
6. Subject must be both motivated and competent to learn to use the Argus II System (by the Investigator's assessment), and willing and able to commit to the study requirements. This includes an understanding of the requirements of the study and acceptance of the time involved in participating;
7. Subject must not suffer from non-ophthalmic serious adverse events (e.g., myocardial infarction, etc.) or from non-curable life threatening conditions (e.g. cancer) at the time of the Baseline visit.

Exclusion Criteria:

1. Ocular diseases or conditions that could prevent the Argus II implant from working (e.g., optic nerve disease, central retinal artery or vein occlusion, history of retinal detachment, trauma, etc.);
2. Evidence of active sub-macular choroidal neovascularization (CNV) in implanted eye;
3. Ocular structures or conditions that could prevent the successful implantation of the Argus II Implant or adequate healing from surgery (e.g. extremely thin conjunctiva; axial length <20.5 mm or > 26 mm; corneal ulcers; abnormalities in the typical curvature of the retina like staphyloma and all causes of significant protrusions or depressions in the area centralis that could compromise the optimal position of the electrode array, active or severe blepharitis, etc.);
4. Ocular diseases or conditions (other than cataracts) that prevent adequate visualization of the inner structures of the eye (e.g., corneal opacity);
5. An Implantable Miniature Telescope in either eye;
6. Pre-disposition to eye rubbing;
7. Any disease or condition that prevents understanding or communication of informed consent, study demands, and testing protocols, including:

   1. cognitive decline including diagnosed forms of dementia and/or progressive neurologic disease,
   2. psychiatric disease including diagnosed forms of depression;
   3. does not speak a principal language associated with the region, and
   4. deafness or selective frequency hearing loss that prevents hearing device alarms and alerts;
8. Pregnant or wish to become pregnant during the course of the study;
9. Participating in another investigational drug or device study that may conflict with the objectives, follow-up or testing of this study;
10. Inability to tolerate general anaesthesia or the recommended antibiotic and steroid regimen associated with the implantation surgery;
11. Conditions likely to limit life to less than 1 year from the time of inclusion.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2015-06; Primary Completion 2019-09 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 1 year
  The number of adverse events in implanted subjects.
Visual function | 1 Year
  The primary effectiveness endpoint of the study is the effect of the Argus II System on monocular (implanted eye) and binocular visual function, as measured by a suite of visual function tests.

CONTACTS AND LOCATIONS:
Overall Officials: Jessy Dorn, PhD, Study Director — Second Sight Medical Products, Inc.
Locations (1):
- Manchester Royal Eye Hospital, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No